CLINICAL TRIAL: NCT01906086
Title: Effects of Legume Consumption on Adiponectin and Inflammatory Markers Among First Degree Relatives of Diabetic Patients
Brief Title: Effects of Legume Consumption on Adiponectin and Inflammatory Markers Among Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Isfahan University of Medical Sciences (Other)
Responsible Party: Principal Investigator, Leila Azadbakht, Isfahan University of Medical Sciences, Isfahan University of Medical Sciences
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Health Services Research
Other Study IDs: legume consumption in adults
Record Dates: First submitted 2013-06-25; First posted 2013-07-23 (Estimated); Last update posted 2014-05-20 (Estimated); Status verified 2014-05

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- legume consumption (Experimental): legume consumption, 4 servings per week, for 6 weeks
  Interventions: Other: nutritional intervention
- healthy dietary recommendations (Active Comparator): no nutritional intervention
  Interventions: Other: life style intervention

INTERVENTIONS:
Other: nutritional intervention
  Arms: legume consumption
Other: life style intervention
  Arms: healthy dietary recommendations

SUMMARY:
The aim of this randomized cross-over study was to determine the effects of legume consumption on adiponectin and inflammatory factors among first degree relatives of diabetic patients

ELIGIBILITY:
Inclusion Criteria:

* age more than 30 years
* no history of chronic diseases
* no use of blood glucose lowering drugs

Exclusion Criteria:

* do not use recommended amounts of legumes
* incidence of chronic diseases during the study
* to start use of blood glucose lowering drugs

Ages: 30 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2012-09; Primary Completion 2013-01 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
high sensitive C reactive protein (mg/l) | 14 weeks
  amounts of hs-CRP

SECONDARY OUTCOMES:
Interleukin-6 (pg/ml) | 14 weeks
  amounts of IL-6
Tumor necrosis factor-α (pg/ml) | 14 weeks
  amounts of TNF-α
Adiponectin (ng/ml) | 14 weeks
  amounts of adiponectin

CONTACTS AND LOCATIONS:
Locations (1):
- Isfahan University of Medical Sciences, Isfahan, Iran